CLINICAL TRIAL: NCT02494544
Title: A Prospective, Multicenter Study to Evaluate Functional Outcome After Knee Replacement
Brief Title: A Multicenter Study to Evaluate Functional Outcome After Knee Replacement
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Decision of investigational team
Sponsor: Restor3D (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Basic Science
Other Study IDs: 12-005
Record Dates: First submitted 2015-05-28; First posted 2015-07-10 (Estimated); Results first posted 2025-10-08 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Osteoarthritis
Keywords: knee implant; knee replacement; total knee replacement
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Site staff that is performing functional testing on subject is blinded to what implant the patient has.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (6):
- ConforMIS iTotal Knee replacement (Active Comparator): iTotal patient-specific knee replacement system
  Interventions: Device: ConforMIS iTotal Knee Replacement
- DePuy total knee replacement (Active Comparator): Off the shelf knee replacement system
  Interventions: Device: Off the Shelf Total Knee Replacement
- Zimmer total knee replacement (Active Comparator): Off the shelf knee replacement system
  Interventions: Device: Off the Shelf Total Knee Replacement
- Biomet total knee replacement (Active Comparator): Off the shelf knee replacement system
  Interventions: Device: Off the Shelf Total Knee Replacement
- Smith & Nephew total knee replacement (Active Comparator): Off the shelf knee replacement system
  Interventions: Device: Off the Shelf Total Knee Replacement
- Stryker total knee replacement (Active Comparator): Off the shelf knee replacement system
  Interventions: Device: Off the Shelf Total Knee Replacement

INTERVENTIONS:
Device: Off the Shelf Total Knee Replacement — A knee replacement system by DePuy, Zimmer, Biomet, Smith & Nephew, or Stryker
  Arms: Biomet total knee replacement; DePuy total knee replacement; Smith & Nephew total knee replacement; Stryker total knee replacement; Zimmer total knee replacement
Device: ConforMIS iTotal Knee Replacement — A knee replacement performed with patient specific implant and surgical jigs.
  Arms: ConforMIS iTotal Knee replacement

SUMMARY:
Patients will be consecutively enrolled by implant. Implant groups will be those who have undergone surgery with either a ConforMIS iTotal® CR TKA or an Off-the- Shelf (OTS) system.

The patient will conduct functional testing and answer questionnaires.

The results will compare the ConforMIS iTotal with an Off the Shelf Knee replacement.

DETAILED DESCRIPTION:
To compare functional and patient reported outcome data for a consecutively enrolled group of subjects who have undergone surgery with either a ConforMIS iTotal® CR TKA or an Off-the- Shelf (OTS) system.The person conducting the functional testing will be blinded to the device implanted. Sites will perform the off-the-shelf total knees conventional instrumentation.

ELIGIBILITY:
Inclusion:

* Clinical condition included in the approved Indications For Use for the iTotal CR
* Osteoarthritis, as confirmed by the investigator's assessment of disease status at screening visit that warrants a TKR procedure. Disease status is assessed by Clinical and Radiographic assessment
* Willingness to participate in the clinical study, to give informed consent and to attend all follow-up visits
* > 18 years of age

Exclusion:

* Subject will require a simultaneous bilateral procedure
* Other lower extremity surgery within 1 year
* Severe (> 15º) fixed valgus or varus deformity
* Severe (> 15º) extension deficit
* Severe instability due to advanced loss of osteochondral structure
* Loss of bone or musculature, osteoporosis, neuromuscular or vascular compromise in the area of the joint to be operated on to an extent that the procedure is unjustified
* Insufficient bone stock on the femoral or tibial surfaces
* Contralateral knee replacement surgery within the past 6 months
* BMI > 40
* Active malignancy (defined as a history of any invasive malignancy - except non-melanoma skin cancer), unless patient has been treated with curative intent and there have been no clinical signs or symptoms of the malignancy for at least 5 years
* Poorly controlled diabetes (defined as HbA1c >7 or surgeon discretion)
* Immunocompromised
* Other physical disability affecting the hips, spine, or contralateral knee that limits function
* Disabling chronic pain with narcotic dependence
* Compromised PCL or collateral ligament
* Prior history of failed implant surgery of the joint to be treated, including Unicompartmental Knee Arthroplasty (UKA), or Bicompartmental Knee Arthroplasty (BKA)
* Prior history of failed high tibial osteotomy (HTO)
* Participation in another clinical study which would confound results
* Inability to complete the protocol in the opinion of the clinical staff due to safety or other reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2015-07-01 (Actual); Primary Completion 2022-11-16 (Actual); Study Completion 2022-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary O'Connor, MD, Principal Investigator — Yale University
Locations (8):
- United States (8):
  - University of California in San Diego, La Jolla, California
  - Sharp Healthcare, San Diego, California
  - Denver-Vail Orthopedics, Parker, Colorado
  - Yale School of Medicine, New Haven, Connecticut
  - Tufts University, Boston, Massachusetts
  - University of Missouri, Columbia, Missouri
  - OrthoNY, Albany, New York
  - The Lindner Center for Research and Education, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: While "Biomet Total Knee Replacement" and "Smith and Nephew Total Knee Replacement" Arms/Groups were listed as possible study groups, no included patients utilized these implant systems. This included patients who failed to meet screening criteria, failed to reach the protocol's required follow-up duration, etc. These arms/groups were only established before the study to represent the possible study groups based on available implant systems on the market.
Period: Overall Study
Arm/Group | ConforMIS iTotal Knee Replacement | DePuy Total Knee Replacement | Zimmer Total Knee Replacement | Biomet Total Knee Replacement | Smith & Nephew Total Knee Replacement | Stryker Total Knee Replacement
Started | 131 | 38 | 19 | 0 | 0 | 26
Completed | 81 | 28 | 19 | 0 | 0 | 19
Not Completed | 50 | 10 | 0 | 0 | 0 | 7

BASELINE CHARACTERISTICS:
Population: Our analysis expected a broader range of off the shelf implants, but no included patients received Biomet or Smith & Nephew Total Knee Replacements.
Groups:
- Total: Total of all reporting groups
Arm/Group | ConforMIS iTotal Knee Replacement | DePuy Total Knee Replacement | Zimmer Total Knee Replacement | Biomet Total Knee Replacement | Smith & Nephew Total Knee Replacement | Stryker Total Knee Replacement | Total
Number analyzed (Participants) | 81 | 28 | 19 | 0 | 0 | 19 | 147
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 42 | 10 | 10 | 0 | 0 | 5 | 67
  >=65 years | 39 | 18 | 9 | 0 | 0 | 14 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.728 (7.482) | 67.321 (6.842) | 63 (8.524) |  |  | 68.105 (6.590) | 65.986 (7.468)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 19 | 13 |  |  | 12 | 89
  Male | 36 | 9 | 6 |  |  | 7 | 58
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 |  |  | 0 | 0
  Asian | 0 | 2 | 0 |  |  | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 |  |  | 0 | 0
  Black or African American | 12 | 6 | 0 |  |  | 2 | 20
  White | 68 | 16 | 19 |  |  | 17 | 120
  More than one race | 0 | 0 | 0 |  |  | 0 | 0
  Unknown or Not Reported | 1 | 4 | 0 |  |  | 0 | 5
Region of Enrollment [Number; unit: participants]
  United States | 73 | 27 | 19 |  |  | 10 | 128
  Germany | 8 | 1 | 0 |  |  | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Functional Activities Subscale Score Within the Knee Society Score (KSS) Measure
Description: Comparing the functional testing differences between iTotal and off the shelf. "Total Functional Activities Score" - a subscale within the Knee Society Score (KSS) with its individual subscale score. The Total Functional Activities Score subscale interprets the functional knee health of each patient via a series of tests such as walking/standing (30 points), standard activities (30 points), advanced activities (25 points), and sports/recreational activities (15 points). Deductions to score are made for factors that limit a patient's mobility, such as needing to use an ambulatory device. The subscale scoring system ranges from 0-100, with higher scores indicating better knee function.
Time Frame: 1 year
Population: Patients that met inclusion criteria and had KSS Total Functional Activities Score.
Measure: Mean (Standard Deviation); unit: Score on a subscale
Arm/Group | ConforMIS iTotal Knee Replacement | DePuy Total Knee Replacement | Zimmer Total Knee Replacement | Biomet Total Knee Replacement | Smith & Nephew Total Knee Replacement | Stryker Total Knee Replacement
Number analyzed (Participants) | 73 | 26 | 18 | 0 | 0 | 15
Score on a subscale
  Baseline Score | 42.34 (16.31) | 40.38 (13.07) | 43.56 (12.38) |  |  | 38.87 (13.53)
  1 Year Score | 77.16 (16.47) | 73.65 (16.99) | 88.94 (6.20) |  |  | 71.20 (23.63)
  Change in Score | 34.82 (21.73) | 33.27 (18.28) | 45.39 (13.18) |  |  | 32.33 (19.21)

2. Secondary Outcome: Patient Satisfaction Subscale Score Within the Knee Society Score (KSS) Measure
Description: Measuring and comparing the differences between iTotal and off the shelf knees with patient reported outcomes. "Patient Satisfaction", a subscale within the Knee Society Score (KSS), was utilized to capture this metric. The Patient Satisfaction subscale combines scores given for certain responses (very satisfied, satisfied, neutral, somewhat dissatisfied, very dissatisfied) across 5 questions. These questions are designed to determine the level of satisfaction a patient has with their implant across both everyday and active activities. This score ranges from 0-40, with higher scores indicating higher levels of patient satisfaction.
Time Frame: 1 year
Population: Patients that met inclusion criteria and had patient satisfaction data were included.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ConforMIS iTotal Knee Replacement | DePuy Total Knee Replacement | Zimmer Total Knee Replacement | Biomet Total Knee Replacement | Smith & Nephew Total Knee Replacement | Stryker Total Knee Replacement
Number analyzed (Participants) | 73 | 26 | 18 | 0 | 0 | 15
score on a scale
  Baseline Score | 12.49 (7.09) | 13.62 (6.50) | 15.67 (7.65) |  |  | 15.50 (6.67)
  1 Year Score | 33.78 (8.28) | 32.00 (7.80) | 37.44 (3.81) |  |  | 32.93 (6.84)
  Change in Score | 21.29 (10.76) | 18.38 (9.63) | 21.78 (8.08) |  |  | 17.73 (8.71)

3. Secondary Outcome: Incidents of Major Procedure-related and Device Related Complications (Including Revision Rates)
Description: All complications were stratified according to clinicaltrials.gov reporting standards and each site labeled each complication as either device-related, non-device-related, procedure-related, and non-procedure-related.
Time Frame: 1 year
Population: No included patients utilized the Biomet or Smith & Nephew total knee replacement systems.
Measure: Number; unit: Patients with Events
Arm/Group | ConforMIS iTotal Knee Replacement | DePuy Total Knee Replacement | Zimmer Total Knee Replacement | Biomet Total Knee Replacement | Smith & Nephew Total Knee Replacement | Stryker Total Knee Replacement
Number analyzed (Participants) | 81 | 28 | 19 | 0 | 0 | 19
Patients with Events
  Major Procedure Related Complications | 12 | 5 | 1 |  |  | 3
  Device Related Complications (including revision) | 1 | 0 | 0 |  |  | 0

ADVERSE EVENTS:
Time Frame: 1 year post-operation.
Description: Adverse event collection followed the definitions given on clinicaltrials.gov
Arm/Group | ConforMIS iTotal Knee Replacement | DePuy Total Knee Replacement | Zimmer Total Knee Replacement | Biomet Total Knee Replacement | Smith & Nephew Total Knee Replacement | Stryker Total Knee Replacement
All-Cause Mortality (participants affected / at risk) | 0/81 | 0/28 | 0/19 | 0/0 | 0/0 | 0/19
Serious Adverse Events (participants affected / at risk) | 13/81 | 6/28 | 2/19 | 0/0 | 0/0 | 0/19
Other Adverse Events (participants affected / at risk) | 26/81 | 7/28 | 1/19 | 0/0 | 0/0 | 7/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ConforMIS iTotal Knee Replacement (N=81) | DePuy Total Knee Replacement (N=28) | Zimmer Total Knee Replacement (N=19) | Biomet Total Knee Replacement (N=0) | Smith & Nephew Total Knee Replacement (N=0) | Stryker Total Knee Replacement (N=19)
SAS (General disorders) | 13 | 6 | 2 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ConforMIS iTotal Knee Replacement (N=81) | DePuy Total Knee Replacement (N=28) | Zimmer Total Knee Replacement (N=19) | Biomet Total Knee Replacement (N=0) | Smith & Nephew Total Knee Replacement (N=0) | Stryker Total Knee Replacement (N=19)
Procedure Related Complication (Injury, poisoning and procedural complications) | 12 (12) | 5 (5) | 1 (1) | NA | NA | 3 (3)
Infection-related Complication (Infections and infestations) | 5 (5) | 0 (0) | 0 (0) | NA | NA | 1 (1)
Wound Complications (General disorders) | 5 (5) | 0 (0) | 0 (0) | NA | NA | 1 (1)
Thrombotic Complications (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | NA | NA | 2 (2)
Pain/Stiffness Complications (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2) | 0 (0) | NA | NA | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-27): https://cdn.clinicaltrials.gov/large-docs/44/NCT02494544/Prot_SAP_000.pdf